CLINICAL TRIAL: NCT02660749
Title: The Effect Of Tramadol, Metamizol and Dexketoprofen Combination On Chronic Pain Development After Heart Surgery
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Tobb University of Economics and Technology (Other)
Responsible Party: Sponsor
Other Study IDs: 2015-PMS-41
Record Dates: First submitted 2016-01-18; First posted 2016-01-21 (Estimated); Last update posted 2016-01-21 (Estimated); Status verified 2015-12

CONDITIONS: Heart Surgery

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Non Coronary Heart Surgery scheduled for the study , in patients with acute postoperative period Use of tramadol retard, metamizol and dekxketoprofen the effects on pain and character has been seen in the chronic phase targeted.

DETAILED DESCRIPTION:
This prospective study analyzed surgical thoracotomy and sternotomy patients treated with analgesic drug when higher than 4 regularly. Clinical parameters include general demographics, preoperative and postoperative clinical examination status, pain scores, neuropathic pain scores, medication side effects, additional analgesic, antiemetic and lacsatif needs, vital functions, chest drains, blood transfusion needs, duration of cardiopulmonary bypass, cross clamp time and anaesthesia time. The screening tests for neuropathic pain is the Douleur Neuropathique 4. Using at postopertative 3.month DN4 questionnaires predict persistent postoperative neuropathic pain.

ELIGIBILITY:
Inclusion Criteria:

* Patients included between 20-70 years
* ASA 1-4
* Euroscore value lower than 7
* Undergoned non coronary heart surgery (minithoracotomy and sternotomy)
* Intensive care has been discharged from the service in 24 hours , with patients given tramadol retard , metamizol, Dexketoprofen on postoperatif first day to discharged from the hospital.

Exclusion Criteria:

* Diabetes mellitus
* Chronic renal failure
* COPD
* Uncontrolled hypertension
* Epilepsy
* Psychiatric disease
* Malignancy
* Patients with a history of cerebrovascular disease
* Patients with ischemia
* Patients suffering from chronic pain and analgesic use
* Patients taking antidepressants and antiepileptic drug
* Off-pump technique used or redo undergo cases
* Ongoing postoperative time thoracic or mediastinal drains more than 48 hours remaining patients, bleeding or patients who received repeated revisions due to infection
* More than 24 hours remaining in intensive care patients
* Patients with long discharge duration 1 week
* Patients who discontinued due to side effects of tramadol may begin after medicines.
* Postoperative wound infection.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Female and male are being participant.
Sampling Method: Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2015-05; Primary Completion 2016-05 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
neuropathic pain assesement by DN4 score after minithoracotomy and sternotomy | outcome measure assessed 3 months after the surgery

CONTACTS AND LOCATIONS:
Overall Officials: H. Evren Eker, Ass Prof, Study Director — Baskent University Department of Anesthesiology